CLINICAL TRIAL: NCT04311255
Title: Comparing the Efficacy and Safety of Ultrasound Guided Supraclavicular Block Combined With Either Intercosto-brachial Nerve Block or pec11block for Creation of Surgical Brachio-basilic Fistula in Chronic Renal Failure Patients on Hemodialysis
Brief Title: Comparing the Efficacy and Safety of Ultrasound Guided Supraclavicular Block Combined With Either Intercostobrachialor Pec 11for Creation of Surgical Brachio-basilic Fistula in Chronic Renal Failure Patients on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Fathy Hefni,MD-EDIC, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FMASU R 25/2019
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Best Regional Nerve Block for Creation of Surgical Brachiobasilic Fistula
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- intercostal group (Active Comparator): group of patient receiving inrercostal nerve block as analgesia
  Interventions: Procedure: regional anesthesia for the upper limb
- pecs group (Active Comparator): group of patient receiving pectoralis nerve block as analgesia
  Interventions: Procedure: regional anesthesia for the upper limb

INTERVENTIONS:
Procedure: regional anesthesia for the upper limb — pecs-II block and intercostal nerve block

SUMMARY:
In our study we are trying to reach to the more efficient us guided peripheral nerve block either intercosto-brachial or PPEC 11 that can be combined with us guided supraclavicular block to effectively anesthetise the surgical site for creation of brachio-basilic fistula as regarding onset of surgical anesthesia, adequacy of intra-operative anesthesia, the need for surgical wound infiltration, duration of postoperative analgesia and the failure rate of the fistulae.

DETAILED DESCRIPTION:
* Type of Study: Randomized Prospective trail
* Study Setting: Ain Shams University Hospitals, Cairo, Egypt
* Study Period: 6 months.

Sampling Method: Patients will be subdivided randomly into two groups :

Group (SI) : 25 ml of bupivacaine 0.5 % for us guided supraclavicular block plus 10 ml of lidocaine 2% for us guided intercostobrachial nerve block.

Group(SP) : 25 ml of bupivacaine 0.5 % for us guided supraclavicular block plus10 ml of lidocaine 2% for us guided PECll block.

Study Procedures:

Following local university ethical committee approval, informed consent will be obtained. Details of the anesthetic technique and the study protocol will be fully explained at the preoperative visit, and written consent will be obtained from each patient before inclusion in the study. The patients has to have normal prothrombin (PT) and partial thromboplastin (PTT) times before the procedure.

In the pre-induction room the patients will be taught how to assess their own pain score using the numerical rating scale (NRS) (0-10; 0 = no pain, 10 = worst imaginable pain) .

On arrival at the operating room, standard monitoring will be established with five lead electrocardiogram, non-invasive blood pressure measurement and pulse oximeter. After insertion of a 20-gauge intravenous cannula in the non operated arm, an intravenous crystalloid solution will be administered. Supplemental oxygen will be supplied through nasal cannula. The oxygen flow will be set at 3 L/ min.

Patients will receive 1-2 md midazolam intravenous as premedication before the block. All blocks will be performed by one of the authors, The patients will be randomly allocated to one of the two groups, either supraclavicular-intercostobrachial group(SI Group) ,or the supraclavicular-Pec 11 group(SP Group) .

The patient in SI Group is placed in a semi-sitting position by elevating the head of bed 45 degrees with the patients head turned to the opposite site to be blocked. The skin of the neck and the upper chest and axilla and medial upper arm will be prepared in an aseptic fashion. Ultrasound examination of the supraclavicular area will be performed using a 38-mm high frequency (9-12 MHz) linear array transducer with the in-plane approach, will receive 25 ml of 0.5% bupivacaine in the supraclavicular area ,then the operated arm will be abducted and externally rotated, and the elbow flexed to 90°. Ultrasound examination of the medial upper arm will be performed using a 38-mm high frequency (9-12 MHz) linear array transducer and the intercosto-brachial nerve is identified and blocked using 10 ml of lidocaine 2% . The patient in SP Group will also have supraclavicular block that will be performed in the same way as the previous group and then patient is placed in the supine position with the arm abducted 90 degrees position to receive Peg 11 lock by injecting 10ml of lidocaine 2% between pectoralis minor and serratus anterior at 3rd rib level using a 38-mm high frequency (9-12 MHz) linear array transducer with the in-plane approach. The sensory and motor blocks will be evaluated every 5 min for 30 min or until blocks will be complete. An adequate surgical anesthesia will be defined as a motor score of ≥1 , with an absence of pinprick sensations in the area of all the four terminal nerves.

The zero time for onset of sensory and motor blocks will be the completion of the LA injection. Sensory block assessment (0, no block 1, loss of sensation of pinprick 2, loss of sensation of touch) will be performed in the innervations of the four nerve areas, radial (radial dorsum of the hand), median (thenar eminence), ulnar (hypothenar eminence),and intercostobrachial (medial upper arm) corresponding to the nerve distributions in the forearm and hand using the pinprick test, and will be compared with the same stimulation on the contra-lateral arm. The degree of motor block will be evaluated by thumb abduction (radial nerve), thumb adduction (ulnar nerve), and thumb opposition (median nerve), using a 3-point scale (0 =normal motor function, 1 = decreased motor strength, 2 = complete motor block). The onset times of the sensory block (the time between the end of the LA injection and the total abolition of the pinprick response) and motor block (time between the end of the LA injection and complete motor block) will be recorded for each nerve. Patients who will not achieve satisfactory levels of anesthesia and will need intraoperative local infiltration will be recorded .Patient in whom the block failed and local infiltration is not enough will receive general anesthesia (propofol 2mg/kg plus fentanyl 1ug/kg and atracurium 0.5mg/kg ) with laryngeal mask airway inserted for mechanical ventilation .

Postoperative pain will be assessed by one of the authors using a visual analog scale (0, no pain; 10, worst pain imaginable). Analgesic for the first complain of pain will be standardized and consisted of 500 mg of oral or intravenous paracetamol given for a pain score of 4 of visual analog scale.The time to first analgesic requirement will be also recorded by the same author.

Heart rate, peripheral oxygen saturation, respiratory rate, and blood pressure will be measured before the supraclavicular block and 5, 10, 20, 30, 45, and 60 min after the block and thereafter every 60 min for 2 h postoperatively. University of Michigan Sedation Scale (UMSS) (1, awake and alert; 2, sedated, responding to verbal stimulus; 3, sedated, responding to strong physical stimulus; 4, not arousable) will be measured first as baseline before the block then at the same time points for measuring vital signs post-block .

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Grade III, age 25-75 years who are scheduled for brachio-basilic AVF.

Exclusion Criteria:

Patients will be excluded if they have infection at the injection site, allergy to local anesthetics, chronic use of opioids, a history of neurological neuromuscular, or severe hepatic or cardiopulmonary disease, a contraindication to regional anesthesia or patient /guardian refusal.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-04-13 (Actual); Primary Completion 2020-05-03 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with adequate block (no need for intraoperative local infiltration), | "through study completion ,an average of one year"
  ratio

SECONDARY OUTCOMES:
onset of surgical anesthesia | "through study completion ,an average of one year"
  time
duration of postoperative analgesia | "through study completion ,an average of one year"
  time
the failure rate of the fistulae. | "through study completion ,an average of one year"
  Ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Unuversity Hospitals, Cairo, Egypt